CLINICAL TRIAL: NCT02985996
Title: Body Compartment PK for New HIV Pre-exposure Prophylaxis Modalities
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Colleen Kelley, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00092488
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-08

CONDITIONS: HIV Infections
Keywords: Preventative Medicine; Infectious Diseases; Sexually Transmitted Diseases
MeSH Terms: conditions — HIV Infections; Communicable Diseases; Sexually Transmitted Diseases | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase I/Pre-Drug (No Intervention): Ten participants will be asked to complete study phase 1. Participants will be asked to provide blood and urine samples and undergo penile, urethral, and rectal swabs. Up to 12 rectal biopsies will be taken.
- Phase II/Genvoya (Experimental): Participants will receive one dose Genvoya. Participants will be asked to provide blood and urine samples and undergo penile, urethral, and rectal swabs. Up to 12 rectal biopsies will be taken.
  Interventions: Drug: Genvoya
- Phase II/Truvada (Experimental): Participants will receive one dose of Truvada. Participants will be asked to provide blood and urine samples and undergo penile, urethral, and rectal swabs. Up to 12 rectal biopsies will be taken.
  Interventions: Drug: Truvada
- Phase III/Genvoya (Experimental): Participants will receive Genvoya once daily for ten days. Participants will be asked to provide blood and urine samples and undergo penile, urethral, and rectal swabs. Up to 12 rectal biopsies will be taken.
  Interventions: Drug: Genvoya
- Phase III/Truvada (Experimental): Participants will receive Truvada once daily for ten days. Participants will be asked to provide blood and urine samples and undergo penile, urethral, and rectal swabs. Up to 12 rectal biopsies will be taken.
  Interventions: Drug: Truvada

INTERVENTIONS:
Drug: Truvada — Truvada is intended for the treatment of HIV-1 infection. Truvada is a combination of emtricitabine 200 mg and tenofovir disoproxil fumarate 300 mg in one tablet.
  Arms: Phase II/Truvada; Phase III/Truvada
Drug: Genvoya — Genvoya is a 1-pill, once-a-day prescription medicine used to treat HIV-1. Genvoya is a combination of 150 mg of elvitegravir, 150 mg of cobicistat, 200 mg of emtricitabine, and 10 mg of tenofovir alafenamid in one tablet.
  Arms: Phase II/Genvoya; Phase III/Genvoya

SUMMARY:
The purpose of this study is to determine the ability of new anti-HIV agents to penetrate different body compartments in HIV negative men who have sex with men and transgender women. These new agents might be considered for pre-exposure prophylaxis regimens in the future. This study will include 90 healthy, HIV-negative men who have sex with men and transgender women who are not taking hormones aged 18-49 years. Participant must be willing to participate in 1 of the 3 study phases, be willing to take Truvada® (PrEP) or Genvoya®, and willing to undergo blood draws, urethral swabs, and rectal biopsy procedures.

DETAILED DESCRIPTION:
Men who have sex with men (MSM) and Transgender women (TGW) who have sex with men continue to be disproportionately affected by HIV. Over 60% of new HIV infections in the US occur among MSM. The majority of HIV infections among MSM and TGW occur through exposure to the rectal mucosa during receptive anal intercourse (RAI). Pre-exposure prophylaxis (PrEP) is a new HIV prevention method that is recommended by CDC and WHO for MSM at risk of HIV infection. PrEP entails taking an anti-HIV medication (Truvada®; tenofovir/emtricitabine) on a daily basis to prevent HIV infection. However, current tenofovir- based regimens have shown to have side effects that researchers are hoping to reduce in newly developed anti-HIV agents. This study is designed to examine the ability of these new agents to penetrate mucosal tissues and potentially prevent HIV infection during RAI exposure for MSM and TGW.

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative man who reports receptive anal sex with another man in the last 6 months
* Male to female transgender women who have sex with men who report receptive anal intercourse with another man in the last 6 months and are not currently taking hormonal therapy or plan to take hormonal therapy for the duration of the study
* Not currently taking PrEP and no plans to initiate during study
* Able to provide informed consent in English
* No plans for relocation in the next 3 months
* Willing to undergo peripheral blood and rectal biopsy sampling
* Willing to use study products as directed
* Willing to abstain from receptive anal intercourse 3 days prior to starting study product and for the duration of the study and for 7 days after any rectal biopsy procedure.

Exclusion Criteria:

* History of inflammatory bowel disease or other inflammatory, infiltrative, infectious or vascular condition involving the lower gastrointestinal tract that, in the judgment of the investigators, may be worsened by study procedures or may significantly distort the anatomy of the distal large bowel
* Significant laboratory abnormalities at baseline visit, including but not limited to:

  1. Hgb ≤ 10 g/dL
  2. PTT > 1.5x ULN or INR > 1.5x ULN
  3. Platelet count <100,000
  4. Creatinine clearance <60
* Any known medical condition that, in the judgment of the investigators, increases the risk of local or systemic complications of endoscopic procedures or pelvic examination, including but not limited to:

  1. Uncontrolled or severe cardiac arrhythmia
  2. Recent major abdominal, cardiothoracic, or neurological surgery
  3. History of uncontrolled bleeding diathesis
  4. History of colonic, rectal, or vaginal perforation, fistula, or malignancy
  5. History or evidence on clinical examination of ulcerative, suppurative, or proliferative lesions of the anorectal or vaginal mucosa, or untreated sexually transmitted disease with mucosal involvement
* Continued need for, or use during the 14 days prior to enrollment, of the following medications:

  1. Aspirin or more than 4 doses of NSAIDs
  2. Warfarin, heparin (low-molecular weight or unfractionated), platelet aggregation inhibitors, or fibrinolytic agents
  3. Any form of rectally administered agent besides products lubricants or douching used for sexual intercourse
* Continued need for, or use during the 90 days prior to enrollment, of the following medications:

  1. Systemic immunomodulatory agents
  2. Supraphysiologic doses of steroids
  3. Experimental medications, vaccines, or biologicals
* Intent to use HIV antiretroviral pre-exposure prophylaxis (PrEP) during the study, outside of the study procedures
* Symptoms of an untreated rectal sexually transmitted infection (e.g. rectal pain, discharge, bleeding, etc.)
* Current use of hormonal therapy
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Kelley, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 24 participants were recruited in Phase II, but only 18 were randomized to either Genvoya or Truvada due to lost to follow up.
  19 participants were recruited in Phase III, but only 16 were randomized to either Genvoya or Truvada due to lost to follow up.
Groups:
- Phase I/Pre-Drug: Participants will be asked to complete study phase 1. Participants will be asked to provide blood and urine samples and undergo penile, urethral, and rectal swabs. Up to 12 rectal biopsies will be taken.
Period: Overall Study
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Started | 5 | 8 | 10 | 7 | 9
Completed | 5 | 7 | 9 | 7 | 9
Not Completed | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I/Pre-Drug: Participants will be asked to provide blood and urine samples and undergo penile, urethral, and rectal swabs. Up to 12 rectal biopsies will be taken.
- Phase II/Truvada: Experimental: Phase II/Truvada Participants will receive one dose of Truvada. Participants will be asked to provide blood and urine samples and undergo penile, urethral, and rectal swabs. Up to 12 rectal biopsies will be taken.
- Total: Total of all reporting groups
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada | Total
Number analyzed (Participants) | 5 | 8 | 10 | 7 | 9 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 8 | 10 | 7 | 9 | 39
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 5 | 8 | 10 | 7 | 9 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 7 | 6 | 4 | 22
  White | 3 | 5 | 2 | 1 | 4 | 15
  More than one race | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 8 | 10 | 7 | 9 | 39

OUTCOME MEASURES:

1. Primary Outcome: Changes in Intracellular Emtricitabine Triphosphate (FTC-TP)
Description: Intracellular emtricitabine triphosphate (FTC-TP) is measured and compared from blood specimen in both arms from baseline to visit 4. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Measure: Median (Full Range); unit: fmol/1000000 PBMC
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 5 | 7 | 9 | 7 | 9
fmol/1000000 PBMC | 0 [0 to 0] | 3380 [2091 to 4320] | 2580 [1531 to 5340] | 6470 [3030 to 15,380] | 7660 [3170 to 10,470]

2. Primary Outcome: Changes in Intracellular Tenofovir Diphosphate (TFV-DP)
Description: Intracellular tenofovir diphosphate (TFV-DP) is measured and compared from blood specimen in both arms from baseline to visit 4. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Measure: Median (Full Range); unit: fmol/1000000 PBMC
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 5 | 7 | 9 | 7 | 9
fmol/1000000 PBMC | 0 [0 to 0] | 213 [111 to 323] | 28 [0 to 32] | 453 [138 to 897] | 80 [0 to 156]

3. Secondary Outcome: Change in Plasma Emtricitabine (FTC) Concentration
Description: Plasma emtricitabine (FTC) concentration is measured from blood specimen. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 5 | 7 | 9 | 7 | 9
ng/mL | 0 [0 to 0] | 30 [12 to 46] | 34 [20 to 206] | 152 [31 to 613] | 280 [66 to 518]

4. Secondary Outcome: Change in Plasma Tenofovir Disoproxil Fumarate (TDF) Concentration
Description: Plasma tenofovir disoproxil fumarate (TDF) concentration is measured from blood specimen. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Measure: Median (Full Range); unit: ng/mL
Groups:
- Phase II/Short Course: Participants will be randomized to receive one dose of Truvada or Genvoya. Participants will be asked to provide blood and urine samples and undergo penile, urethral, and rectal swabs. Up to 12 rectal biopsies will be taken.
  Truvada: Truvada is intended for the treatment of HIV-1 infection. Truvada is a combination of emtricitabine 200 mg and tenofovir disoproxil fumarate 300 mg in one tablet.
  Genvoya: Genvoya is a 1-pill, once-a-day prescription medicine used to treat HIV-1. Genvoya is a combination of 150 mg of elvitegravir, 150 mg of cobicistat, 200 mg of emtricitabine, and 10 mg of tenofovir alafenamid in one tablet.
- Phase III/Steady State: Participants will be randomized to receive Truvada or Genvoya to be taken once daily for ten days. Participants will be asked to provide blood and urine samples and undergo penile, urethral, and rectal swabs. Up to 12 rectal biopsies will be taken.
  Truvada: Truvada is intended for the treatment of HIV-1 infection. Truvada is a combination of emtricitabine 200 mg and tenofovir disoproxil fumarate 300 mg in one tablet.
  Genvoya: Genvoya is a 1-pill, once-a-day prescription medicine used to treat HIV-1. Genvoya is a combination of 150 mg of elvitegravir, 150 mg of cobicistat, 200 mg of emtricitabine, and 10 mg of tenofovir alafenamid in one tablet.
Arm/Group | Phase I/Pre-Drug | Phase II/Short Course | Phase III/Steady State | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 5 | 7 | 9 | 7 | 9
ng/mL | 0 [0 to 0] | 0 [0 to 0] | 28 [20 to 59] | 0 [0 to 0] | 59 [38 to 89]

5. Secondary Outcome: Change in Plasma Tenofovir Alafenamide (TAF) Concentration
Description: Plasma tenofovir alafenamide (TAF) concentration is measured from blood specimen. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Population: TAF was not measured, only the metabolite TFV was measured
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Change in Plasma Elvitegravir (EVG) Concentration
Description: Plasma elvitegravir (EVG) concentration is measured from blood specimen. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 5 | 7 | 9 | 7 | 9
ng/mL | 0 [0 to 0] | 102 [0 to 295] | 0 [0 to 0] | 384 [99 to 705] | 0 [0 to 0]

7. Secondary Outcome: Change in Rectal Emtricitabine (FTC) Concentration
Description: Emtricitabine (FTC) concentration is measured from rectal secretion specimen. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Measure: Median (Full Range); unit: ng/swab
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 5 | 7 | 9 | 7 | 9
ng/swab | 0 [0 to 0] | 288 [0 to 42,450] | 419 [64 to 6935] | 371 [0 to 3830] | 109 [0 to 3900]

8. Secondary Outcome: Change in Rectal Tenofovir Disoproxil Fumarate (TDF) Concentration
Description: Tenofovir disoproxil fumarate (TDF), concentration is measured from rectal secretion specimen. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Measure: Median (Full Range); unit: ng/swab
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 5 | 7 | 9 | 7 | 9
ng/swab | 0 [0 to 0] | 58 [0 to 1195] | 45 [0 to 263] | 533 [0 to 18,400] | 1325 [0 to 6145]

9. Secondary Outcome: Change in Rectal Tenofovir Alafenamide (TAF) Concentration
Description: Tenofovir alafenamide (TAF) concentration is measured from rectal secretion specimen. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Population: The study didn't measure TAF, only the metabolite TFV
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Change in Rectal Elvitegravir (EVG) Concentration
Description: Elvitegravir (EVG) concentration is measured from rectal secretion specimen. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Measure: Median (Full Range); unit: ng/swab
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 5 | 7 | 9 | 7 | 9
ng/swab | 0 [0 to 0] | 405 [55 to 7975] | 0 [0 to 0] | 219 [0 to 54,100] | 0 [0 to 0]

11. Secondary Outcome: Change in Intracellular Tenofovir Alafenamide (TAF) Concentration in Peripheral Blood Mononuclear Cells (PBMCs)
Description: Intracellular tenofovir alafenamide (TAF) concentration is measured from isolated PBMCs collected via blood draw. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Population: The study didn't measure TAF, only the metabolite TFV
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Change in Intracellular Elvitegravir (EVG) Concentration in Peripheral Blood Mononuclear Cells (PBMCs)
Description: Intracellular elvitegravir (EVG) concentration is measured from isolated PBMCs collected via blood draw. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Population: EVG is very difficult to measure intracellularly, therefore the study only measured plasma or extracellular concentrations.
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Change in Intracellular Emtricitabine (FTC) Concentration in Rectal Tissue
Description: Tissue emtricitabine (FTC) concentration is measured from rectal biopsies and isolated cells. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Measure: Median (Full Range); unit: fmol/mg tissue
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 5 | 7 | 9 | 7 | 9
fmol/mg tissue | 0 [0 to 0] | 0 [0 to 11] | 0 [0 to 51] | 27 [0 to 79] | 41 [0 to 110]

14. Secondary Outcome: Change in Intracellular Tenofovir (TFV) Concentration in Rectal Tissue
Description: Intracellular tenofovir (TFV) Concentration in Rectal Tissue is measured from rectal biopsies and isolated cells. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Measure: Median (Full Range); unit: fmol/mg tissue
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 5 | 7 | 9 | 7 | 9
fmol/mg tissue | 0 [0 to 0] | 17 [0 to 65] | 11 [0 to 74] | 0 [0 to 102] | 0 [0 to 17]

15. Secondary Outcome: Change in Tenofovir Alafenamide (TAF) Concentration in Rectal Tissue
Description: Tissue tenofovir alafenamide (TAF) concentration is measured from rectal biopsies and isolated cells. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Population: The study didn't measure TAF, only the metabolite TFV
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Change in Elvitegravir (EVG) Concentration in Rectal Tissue
Description: Tissue elvitegravir (EVG) concentration is measured from rectal biopsies and isolated cells. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Measure: Median (Full Range); unit: ng/mg tissue
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 5 | 7 | 9 | 7 | 9
ng/mg tissue | 0 [0 to 0] | 2.7 [1.2 to 9.8] | 0 [0 to 0] | 6.8 [4.5 to 11.1] | 0 [0 to 0]

17. Secondary Outcome: Change in Emtricitabine (FTC) Concentration in Penile Secretions
Description: Emtricitabine (FTC) concentrations is measured from urethral and penile specimen. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Measure: Median (Full Range); unit: ng/swab
Arm/Group | Phase I/Pre-Drug | Phase II/Short Course | Phase III/Steady State | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 5 | 7 | 9 | 7 | 9
ng/swab | 0 [0 to 0] | 32 [0 to 77] | 30 [0 to 406] | 175 [0 to 1775] | 54 [0 to 9685]

18. Secondary Outcome: Change in Tenofovir Disoproxil Fumarate (TDF) Concentration in Penile Secretions
Description: Tenofovir disoproxil fumarate (TDF) concentrations is measured from urethral and penile specimen. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Measure: Median (Full Range); unit: ng/swab
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 5 | 7 | 9 | 7 | 9
ng/swab | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 385] | 0 [0 to 30] | 17 [0 to 818]

19. Secondary Outcome: Change in Tenofovir Alafenamide (TAF) Concentration in Penile Secretions
Description: Tenofovir alafenamide (TAF) concentrations is measured from urethral and penile specimen. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Population: The study did not measure TAF, only the metabolite TFV
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Change in Elvitegravir (EVG) Concentration in Penile Secretions
Description: Elvitegravir (EVG) concentrations is measured from urethral and penile specimen. For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Baseline, Visit 4 (Up to ten days post drug)
Measure: Median (Full Range); unit: ng/swab
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 5 | 7 | 9 | 7 | 9
ng/swab | 0 [0 to 0] | 0 [0 to 28] | 0 [0 to 0] | 0 [0 to 12] | 0 [0 to 0]

21. Secondary Outcome: PrEP Efficacy as Measured by Inhibition of in Vitro Infection of Rectal Biopsies to HIV
Description: Rectal biopsies will be subjected to in vitro infection with HIV to test for changes in susceptibility to virus infection. Concentrations of cumulative p24 production in supernatants following in vitro infection of rectal biopsies correlate with viral infection and replication in rectal biopsies. Therefore, lower concentrations of p24 production in biopsies collected from men receiving PrEP compared to controls indicates a potential greater protection from infection and potential increased PrEP efficacy.
  For the pharmacokinetic analysis, values reported as "Below the Limit of Quantification" (BLOQ) are assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
Time Frame: Up to 10 months post-baseline
Measure: Median (Full Range); unit: ng p24
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
Number analyzed (Participants) | 5 | 7 | 9 | 7 | 9
ng p24 | 740 [271 to 2319] | 225 [128 to 535] | 298 [224 to 381] | 348 [159 to 504] | 327 [94 to 465]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Phase I/Pre-Drug | Phase II/Genvoya | Phase II/Truvada | Phase III/Genvoya | Phase III/Truvada
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/8 | 0/10 | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/8 | 0/10 | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 0/5 | 0/8 | 0/10 | 0/7 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT02985996/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT02985996/SAP_001.pdf